CLINICAL TRIAL: NCT07308769
Title: A Prospective, Open-Label, Randomized, Interventional Study to Evaluate the Efficacy and Tolerability of Sucrosomial® Iron vs Ferric Maltol in Iron Deficient Women
Brief Title: Efficacy and Tolerability of Sucrosomial® Iron vs Ferric Maltol in Iron Deficient Women
Acronym: SID-WOMEN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Pharmanutra S.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SID-WOMEN; 2025-522004-24-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-17; First posted 2025-12-30 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Anemia; Iron Deficiency Anemia (IDA)
Keywords: Iron Deficiency; Iron Deficiency Anemia; Mild to Moderate Anemia; anemia in women
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency; Iron Deficiencies | interventions — ferric maltol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sucrosomial® Iron (Experimental): Participants will receive dietary supplement Sucrosomial® Iron (Sideral® Forte) for 12 weeks.
  The dose consists of 60 mg/day of elemental iron (two capsules of Sideral® Forte per day), taken orally on an empty stomach (1 hour before or 2 hours after meals).
  Interventions: Dietary Supplement: Sucrosomial® Iron (Sideral® Forte)
- Ferric Maltol (Active Comparator): Participants in this arm will receive Ferric Maltol (Feraccru®) for 12 weeks. The dose consists of 60 mg/day of ferric maltol (two capsules of Feraccru® per day), taken orally on an empty stomach (1 hour before or 2 hours after meals).
  Interventions: Drug: Ferric Maltol (Feraccru®)

INTERVENTIONS:
Dietary Supplement: Sucrosomial® Iron (Sideral® Forte) — Sucrosomial® Iron (Sideral® Forte), 30 mg elemental iron per capsule
  Arms: Sucrosomial® Iron
Drug: Ferric Maltol (Feraccru®) — Ferric Maltol (Feraccru®), 30 mg elemental iron per capsule
  Arms: Ferric Maltol

SUMMARY:
This study aims to compare two oral iron treatments, Sucrosomial® Iron and Ferric Maltol, in women with mild to moderate iron deficiency anemia. Many patients experience gastrointestinal side effects or poor tolerability with traditional iron supplements, which may limit adherence. Participants will be randomly assigned to receive either Sucrosomial® Iron or Ferric Maltol for 12 weeks. The primary objective is to determine whether Sucrosomial® Iron is as effective as Ferric Maltol in normalizing hemoglobin levels.

DETAILED DESCRIPTION:
This prospective, randomized, open-label, two-arm study evaluates whether Sucrosomial® Iron is non-inferior to Ferric Maltol in normalizing hemoglobin levels over 12 weeks in women with mild to moderate iron deficiency anemia. A total of 146 participants will be randomized 1:1 to receive either Sucrosomial® Iron or Ferric Maltol.

The primary endpoint is hemoglobin normalization at Week 12. Secondary endpoints include changes in iron parameters (serum iron, ferritin, transferrin saturation), fatigue improvement using the FACIT-Fatigue Scale, and assessment of tolerability (adverse events, discontinuations). The study includes a screening phase and follow-up visits at Weeks 4, 6, 8, and 12 for safety monitoring, laboratory assessments, and evaluation of treatment compliance.

ELIGIBILITY:
Inclusion Criteria:

* Female participants ≥ 18 years
* Mild anemia (11.0 ≤ Hb < 12 g/dL) or moderate anemia (8.0 < Hb < 11 g/dL)
* Signed informed consent

Exclusion Criteria:

* Use of iron-containing drugs or supplements within 1 month prior to screening
* Psychiatric disorders interfering with consent or compliance
* Active cancer (except fibroids and polyps)
* Pregnant or breastfeeding women
* Participation in another interventional study
* History of poor adherence or inability to comply
* Use of erythropoietin within 3 months prior to screening
* Need for blood transfusion or IV iron (per investigator judgment)
* Severe active IBD (HBI > 16 for Crohn; CAI > 12 for ulcerative colitis)
* Previous bariatric surgery
* Alcohol abuse
* Hemochromatosis or iron overload syndromes
* Hereditary anemias (including thalassemia)
* Known hypersensitivity to study product ingredients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin normalization at week 12 | Week 12 (End of Treatment)
  Proportion of participants achieving hemoglobin ≥ 12 g/dL after 12 weeks of treatment.

SECONDARY OUTCOMES:
Hemoglobin normalization at intermediate timepoints (Week 6 and Week 8) | Week 6 and Week 8
  Proportion of participants who achieve hemoglobin normalization (Hb ≥ 12 g/dL) at Week 6 and Week 8.
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 to Week 12
  Number and proportion of participants experiencing any AEs or SAEs during the study period, assessed at each visit.
Withdrawals due to adverse events | Day 1 to Week 12
  Number of participants who withdraw from the study because of an adverse event.
Treatment discontinuation due to intolerable side effects | Day 1 to Week 12
  Number of participants who discontinue study treatment due to intolerable side effects.
Normalization of iron status markers | Baseline to Week 12
  Proportion of participants achieving normalization of iron parameters: serum iron, ferritin, transferrin saturation (TSAT).
Change from baseline in FACIT-Fatigue Scale (v4.0) | Day 1, Week 4, Week 6, Week 8, Week 12
  Change from baseline in fatigue symptoms using the FACIT-Fatigue Scale v4.0. Higher scores indicate improvement.
Change in hemoglobin levels from baseline at each study visit | Baseline to Week 12 (with assessments at Week 6 and Week 8)
  Mean change in hemoglobin concentration from baseline at each study visit.
Hemoglobin variation in participants with chronic inflammation (CRP-based Subgroups) | Baseline to Week 12
  Change in hemoglobin levels from baseline in participants stratified by CRP category. CRP values categorized as follows: Normal (CRP < 0.3 mg/dl); Normal or minorelevation (0.3 ≤ CRP < 1.0 mg/dl); Moderate elevation (1.0 ≤ CRP ≤ 10.0 mg/dl); Marked elevation (CRP > 10.0 mg/dl).
Acceptability / discontinuation due to taste | Day 1 to Week 12
  Proportion of participants refusing or discontinuing the study treatment due to taste.

CONTACTS AND LOCATIONS:
Locations (7):
- Spain (7):
  - Hospital Quironsalud Barcelona, Barcelona
  - Hospital Universitari Dexeus Grupo Quironsalud, Barcelona
  - Hospital Universitari Sagrat Cor, Barcelona
  - Hospital Quironsalud Malaga, Málaga
  - Hospital Quironsalud Malága, Málaga
  - Hospital Universitari General De Catalunya, Sant Cugat del Vallès
  - Hospital Quironsalud Zaragoza, Zaragoza